CLINICAL TRIAL: NCT01313936
Title: Pilot Study of High-Dose 131I-MIBG Therapy Combined With Vincristine and Five Days of Irinotecan for Resistant/Relapsed High-Risk Neuroblastoma
Brief Title: High-Dose 131I-MIBG Therapy Combined With Vincristine and Five Days of Irinotecan for Resistant/Relapsed Neuroblastoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Thrasher Research Fund (Other)
Responsible Party: Principal Investigator, Steven Dubois, Assistant Professor of Pediatrics, University of California, San Francisco
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MIBG Irino
Record Dates: First submitted 2011-03-10; First posted 2011-03-14 (Estimated); Results first posted 2015-08-07 (Estimated); Last update posted 2019-04-29 (Actual); Status verified 2019-01

CONDITIONS: Neuroblastoma
Keywords: Neuroblastoma; MIBG; 131I-MIBG; Irinotecan; Vincristine; Resistant; Relapsed; Treatment; UCSF; Pediatric; Oncology
MeSH Terms: conditions — Neuroblastoma; Recurrence; Neoplasms | interventions — 3-Iodobenzylguanidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 15 mCi/kg of 131I-MIBG (Experimental): The first cohort for safety will be 3-6 patients treated with vincristine and irinotecan and 15 mCi/kg of 131I-MIBG.
  Interventions: Drug: Metaiodobenzylguanidine (MIBG)
- 18 mCi/kg of 131I-MIBG (Experimental): The second cohort will be 3-6 patients at the same doses of vincristine and irinotecan and 18 mCi/kg of 131I-MIBG.
  Interventions: Drug: Metaiodobenzylguanidine (MIBG)

INTERVENTIONS:
Drug: Metaiodobenzylguanidine (MIBG) — Chemotherapy will be given over 5 days for each course, with a single dose of 131I-MIBG on the second day of irinotecan. A total course will be defined as 42 days, or longer if hematopoietic recovery to eligibility criteria occurs after day 42.
  Other Names: 131I-MIBG

SUMMARY:
This is a pilot study to determine whether doses of 15 mCi/kg and 18 mCi/kg of 131I-MIBG are tolerable when given with irinotecan/vincristine on a one week schedule to children and young adults with high-risk refractory/relapsed neuroblastoma.

DETAILED DESCRIPTION:
131I-metaiodobenzylguanidine (131I-MIBG) is an active therapy in patients with widely metastatic, treatment-resistant neuroblastoma, where response rates are 20-40% at doses (> 15mCi/kg) requiring stem cell rescue. Irinotecan is a topoisomerase I inhibitor with single-agent chemotherapeutic activity against neuroblastoma and other pediatric solid tumors in phase I and II clinical trials. With more protracted schedules (e.g. daily for 5 days/week x 2 weeks), the major dose-limiting toxicity is diarrhea. With shorter schedules, myelosuppression becomes dose-limiting. In adult solid tumors, irinotecan has been an effective radiosensitizer and is currently being evaluated by the Children's Oncology Group for this purpose in rhabdomyosarcoma protocols incorporating external beam radiotherapy.

Compared to single-agent 131I-MIBG, the combination of topotecan (a related camptothecin) and 131I-MIBG demonstrated superior pre-clinical activity in mouse xenograft models of neuroblastoma. This combination had no unexpected toxicities in a pilot clinical study. We have completed a clinical trial of vincristine, irinotecan, 131I-MIBG that utilized irinotecan on a protracted schedule (5 days per week x 2 weeks). The rationale for this schedule was to provide a greater degree of overlap between the radiation sensitizer (irinotecan) and the radiation exposure provided following 131I-MIBG infusion. This combination was shown to be tolerable at doses up to 18 mCi/kg 131I-MIBG. However, more patients experienced grade 2 and 3 diarrhea than would be customary with the dose and schedule of irinotecan used in that trial. It is therefore of interest to determine whether this combination of irinotecan, vincristine, and 131I-MIBG will be better tolerated using irinotecan at higher doses in a shorter schedule. The current standard schedule in Children's Oncology Group protocols for the combination of vincristine, irinotecan is now a higher dose in five, rather than 10 days. In the current pilot study, we will evaluate the tolerability and anti-tumor activity of this combination using irinotecan given once daily for 5 days only. Two 131I-MIBG dose levels will be evaluated. This study will provide the basis for a future randomized trial.

ELIGIBILITY:
Inclusion Criteria:

* Age: Patients must be >1 year and < 30 years of age when registered on study.
* Diagnosis: Patients must have a diagnosis of neuroblastoma either by histologic verification of neuroblastoma and/or demonstration of tumor cells in the bone marrow with increased urinary catecholamines.
* Disease status: Patients must have high-risk neuroblastoma with at least ONE of the following:

  1. Recurrent/progressive disease at any time. Biopsy not required, even if partial response to intervening therapy except in patients with only one site of MIBG-avid disease that has been radiated within the preceding two months. Such patients require biopsy confirmation of residual active disease, with positive bone marrow biopsy being adequate confirmation of residual active disease.
  2. Refractory disease (i.e. less than a partial response to frontline therapy, including a minimum of 4 cycles of induction chemotherapy). No biopsy is required for eligibility for this study.
  3. Persistent disease after at least a partial response to frontline therapy (i.e. patient has had at least a partial response to frontline therapy but still has residual disease by MIBG scan, CT/MRI, or bone marrow). Patients in this category are REQUIRED to have a biopsy (bone marrow biopsy included) of at least one residual site demonstrating viable neuroblastoma.
* 131I-MIBG Uptake: Patients must have evidence of MIBG uptake into tumor at ≥ one site within 4 weeks prior to entry on study and subsequent to any intervening therapy.
* Hematopoietic stem cells: Patients must have an adequate unpurged peripheral blood hematopoietic stem cell product, with a minimum of 2 X 106 CD34+ cells/kg available. Having a back-up of 2.0 x 106 viable CD34+ cells/kg unpurged PBSC is recommended but not required. The use of purged stem cells or autologous bone marrow as donor source is not allowed. The use of PBSC from an identical twin is allowed.
* Performance and life expectancy: Must have a life expectancy of at least 6 weeks and a Lansky or Karnofsky score of at least 60.
* Prior therapy: Patients must have fully recovered from the acute toxic effects of all prior chemotherapy, immunotherapy, or radiotherapy prior to entering this study.

  1. Myelosuppressive chemotherapy and/or biologics: Patients are not required to complete re-induction chemotherapy prior to study entry following relapse. Last dose of any myelosuppressive or biologic therapy was given at least 2 weeks before the start date for irinotecan on this protocol.
  2. Radiation: Patients must not have received radiation for a minimum of two weeks prior to study entry. Patients who received radiation to the only site of MIBG-avid disease within two months of study entry require biopsy confirmation of residual active disease, with positive bone marrow biopsy being adequate confirmation of residual active disease. A minimum of 3 months is required following prior large field radiation therapy (i.e. craniospinal therapy, total lung, > 50% marrow space). Patients are excluded if they have received whole abdominal radiation or TBI (total body irradiation).
  3. Stem Cell Transplant (SCT): Patients are eligible three months after autologous stem cell transplant. Patients status post-allogeneic stem cell transplant are excluded. Must meet adequate bone marrow function definition (see organ function requirements, below) post-myeloablative therapy.
  4. Prior 131I-MIBG therapy: Patients may have received prior MIBG therapy, though cumulative lifetime dose should not exceed 18 mCi/kg prior to study entry. Patients must not have received MIBG in combination with irinotecan. For patients previously treated with MIBG, at least 6 months must have elapsed since last MIBG therapy.
  5. Growth factor(s): All cytokines or hematopoietic growth factors must be discontinued a minimum of 7 days prior to the start date for irinotecan on this protocol.
  6. Prior irinotecan and vincristine therapy: are allowed, subject to recovery of adequate bone marrow function as specified in the protocol.
* Concomitant Therapy Restrictions: Patients must not be receiving any other anti-cancer agents or radiotherapy at the time of study entry or while on study. Enzyme-inducing anticonvulsants (phenobarbital, phenytoin, carbamazepine) must not be used as these may interfere with irinotecan metabolism. Non-enzyme inducing anticonvulsants (Keppra, etc.) can be used after discussion with study chair. The use of high dose dexamethasone and the use of aprepitant as antiemetics is not recommended due to effects on irinotecan metabolism.
* Hematologic function: a. ANC: > 750/uL (no hematopoietic growth factors within 7 days of the start date for irinotecan on this protocol) b. Platelet count: > 50,000/µl, transfusion independent (defined as no platelet transfusion for one week).

  c. These criteria must be met by all patients, regardless of bone marrow involvement with tumor.
* Renal function: a. Glomerular Filtration Rate (GFR) or 12-24hr Creatinine Clearance >= 60 ml/min/1.73 m², OR b. Age-adjusted serum creatinine < 1.5 x normal for age (see below):

Age Maximum Serum Creatinine (mg/dL) < 5 years 0.8 > 5 and < 10 years 1.0 > 10 and < 15 years 1.2 > 15 years 1.5

* Liver function:a. Total bilirubin <= 1.5 x normal for age, and b. SGPT (ALT) and SGOT (AST) < 3 x upper limit of normal
* Cardiac function: Normal ejection fraction (>=55%) documented by either echocardiogram or radionuclide MUGA evaluation OR normal fractional shortening (>= 27%) documented by echocardiogram.
* Lung function: Normal lung function with no dyspnea at rest, exercise intolerance, pleural effusion or oxygen requirement.
* Reproductive function: All post-menarchal females must have a negative urine or serum beta-HCG. Males and females of reproductive age and childbearing potential must use effective contraception for the duration of their participation.
* Coexisting medical conditions: Patients with other ongoing serious medical issues must be approved by the study chair prior to registration.

Exclusion Criteria:

* Pregnant or lactating.
* Patients status post-ALLOGENEIC stem cell transplant are NOT eligible.
* Patients who, in the opinion of the investigator, may not be able to comply with the safety monitoring requirements of the study.
* Patients with disease of any major organ system that would compromise their ability to withstand therapy.
* Patients who are on hemodialysis.
* Patients with a documented allergy to 3rd generation cephalosporins.
* Patients must not have active diarrhea (defined as > Grade 2 per CTCAE v4 [ Grade 2 = increase of 4-6 stools/day over baseline] ).
* Patients with an active or uncontrolled infection, including C. difficile, of > grade 3 per CTCAE v4. Patients on prolonged antifungal therapy are eligible if they are culture and biopsy negative in suspected radiographic lesions and meet other organ function criteria.
* Patients and/or families who are physically and psychologically unable to cooperate with the radiation safety isolation.
* Patients who have received prior total body or whole abdominal radiation.
* Patients who have received prior 131I-MIBG therapy in combination with irinotecan.

Ages: 1 Year to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 32 (Actual)
Dates: Start 2011-03; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven DuBois, M.D., Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 15 mCi/kg of 131I-MIBG | 18 mCi/kg of 131I-MIBG
Started | 6 | 26
Completed | 6 | 26
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 15 mCi/kg of 131I-MIBG | 18 mCi/kg of 131I-MIBG | Total
Number analyzed (Participants) | 6 | 26 | 32
Age, Continuous [Mean (Full Range); unit: years] | 12.5 [4 to 23] | 6 [2 to 30] | 6 [2 to 30]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 9 | 11
  Male | 4 | 17 | 21
Region of Enrollment [Number; unit: participants]
  United States | 6 | 26 | 32

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose-limiting Toxicity as a Measure of Tolerability
Description: To determine whether doses of 15 mCi/kg and 18 mCi/kg of 131I-MIBG are tolerable when given with irinotecan/vincristine on a 5-day schedule to children and young adults with high-risk refractory/relapsed neuroblastoma.
Time Frame: 6 weeks
Measure: Number; unit: participants with DLT
Arm/Group | 15 mCi/kg of 131I-MIBG | 18 mCi/kg of 131I-MIBG
Number analyzed (Participants) | 6 | 26
participants with DLT | 0 | 0

2. Secondary Outcome: Therapeutic Response Rate
Description: Therapeutic response rate to regimen according to the NANT modified-version of the International Neuroblastoma Response Criteria.
Time Frame: 6 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | 15 mCi/kg of 131I-MIBG | 18 mCi/kg of 131I-MIBG
Number analyzed (Participants) | 6 | 26
Participants | 3 | 6

3. Secondary Outcome: Changes in Diarrhea
Description: Rate of protocol associated diarrhea according to UGT1A1 genotype.
Time Frame: One year
Measure: Count of Participants; unit: Participants
Groups:
- Homozygous Wildtype: Wildtype population, no UGT1A1 polymorphisms
- Heterozygous UGT1A1*28 Genotype: Population Heterozygous for UGT1A1*28 polymorphisms
- Homozygous UGT1A1*28 Genotype: Population homozygous UGT1A1*28 genotype polymorphisms
Arm/Group | Homozygous Wildtype | Heterozygous UGT1A1*28 Genotype | Homozygous UGT1A1*28 Genotype
Number analyzed (Participants) | 11 | 8 | 5
Participants
  Diarrhoea (any grade) | 8 | 5 | 4
  Diarrhoea (> grade 2) | 2 | 0 | 0

4. Secondary Outcome: Changes in Standardized Uptake Values on FDG-PET Scans
Description: To describe changes in standardized uptake values (SUVs) obtained by 18FDG-PET scan at study entry and in response to one cycle of protocol therapy.
Time Frame: One year
Population: No PET scans were performed during this trial.
Arm/Group | 15 mCi/kg of 131I-MIBG | 18 mCi/kg of 131I-MIBG
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected over the 6-week observation period.
Description: Adverse events were based upon CTCAE.
Arm/Group | 15 mCi/kg of 131I-MIBG | 18 mCi/kg of 131I-MIBG
Serious Adverse Events (participants affected / at risk) | 0/6 | 2/26
Other Adverse Events (participants affected / at risk) | 0/6 | 2/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 15 mCi/kg of 131I-MIBG (N=6) | 18 mCi/kg of 131I-MIBG (N=26)
dehydration (General disorders) | 0 | 2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 15 mCi/kg of 131I-MIBG (N=6) | 18 mCi/kg of 131I-MIBG (N=26)
Diarrhea (Gastrointestinal disorders) | 0 | 2 — Only grade 3 reported

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No